CLINICAL TRIAL: NCT01643811
Title: Effect of Gastrectomy and Anastomosis on Chronic Metabolic Disease Such as Diabetes and Hypertension in Early Gastric Cancer Patients
Brief Title: Effect of Gastrectomy and Anastomosis on Diabetes and Hypertension in Early Gastric Cancer Patients
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Keun Won Ryu, Principal Investigator, National Cancer Center, Korea
Other Study IDs: 1210552-1
Record Dates: First submitted 2012-07-11; First posted 2012-07-18 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Early Gastric Cancer
Keywords: early gastric cancer, diabetes, hypertension
MeSH Terms: conditions — Stomach Neoplasms; Diabetes Mellitus; Hypertension | interventions — Gastrectomy; Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Gastrectomy: Patients who underwent gastrectomy for early gastric cancer
  Interventions: Procedure: gastrectomy
- Endoscopic submucosal dissection: Patients who underwent endoscopic submucosal dissection for early gastric cancer
  Interventions: Procedure: Endoscopic submucosal dissection

INTERVENTIONS:
Procedure: gastrectomy — subtotal gastrectomy with gastroduodenostomy or loop gastrojejunostomy or Roux Y gastrojejunostomy total gastrectomy with Roux Y esophagojejunostomy
  Groups: Gastrectomy
Procedure: Endoscopic submucosal dissection — endoscopic submucosal dissection
  Groups: Endoscopic submucosal dissection

SUMMARY:
The purpose of this study is to determine whether the extent of gastrectomy and anastomosis type affect chronic metabolic disease such as diabetes and hypertension in early gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary gastric adenocarcinoma
* clinical stage Ia or Ib examined with endoscopy, endoscopic ultrasound, and computed tomography
* aged 20-80 year old,
* performance status (PS) of 0 or 1 on Eastern Cooperative Oncology Group (ECOG) scale
* diagnosed as diabetes or hypertension
* patients planning to undergo gastrectomy or endoscopic submucosal dissection
* written informed consent

Exclusion Criteria:

* having high risk for operation such as severe heart disease, severe respiratory disease
* pregnant
* previous abdominal surgery or radiation therapy
* proven more advanced disease than pathological stage II requiring adjuvant chemotherapy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed as early gastric cancer
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2012-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who quit previous medication for diabetes because of improved disease | 5 year after operation
  proportion of patients who quit their previous medication for diabetes because of improved disease after operation among all patients who underwent gastrectomy for early gastric cancer with diabetes.
Proportion of patients who quit previous medication for hypertension because of improved disease | 5 years after operation
  Proportion of patients who quit previous medication for hypertension because of improved disease among the patients who diagnosed as early gastric cancer and hypertension

SECONDARY OUTCOMES:
difference of proportion of patients who quit previous medication for diabetes between patients who underwent subtotal gastrectomy and those who underwent total gastrectomy | 5 years after operation
  difference of proportion of patients who quit previous medication for diabetes between patients who underwent subtotal gastrectomy and those who underwent total gastrectomy
difference of proportion of patients who quit previous medication for diabetes according to anastomosis | 5 year after operation
  difference of proportion of patients who quit previous medication for diabetes among patients who underwent gastroduodenostomy and loop gastrojejunostomy and Roux-Y gastrojejunostomy
difference of proportion of patients who quit previous medication for hypertension between patients who underwent subtotal gastrectomy and those who underwent total gastrectomy | 5 years after operation
  difference of proportion of patients who quit previous medication for hypertension between patients who underwent subtotal gastrectomy and those who underwent total gastrectomy
difference of proportion of patients who quit previous medication for hypertension according to anastomosis | 5 years after operation
  difference of proportion of patients who quit previous medication for hypertension among patients who underwent gastroduodenostomy and loop gastrojejunostomy and Roux-Y gastrojejunostomy
difference of serum levels of c-peptide, Ghrelin, GIP, GLP-1, glucagon, insulin between before and after operation | 1 years after operation
  difference of serum levels of c-peptide, Ghrelin, GIP, GLP-1, glucagon, insulin between before and after operation in patients with diabetes

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang, Kyeonggi-do, South Korea